CLINICAL TRIAL: NCT05466097
Title: Development of Polygenic Risk Score to Predict the Efficacy of Weight Loss Intervention in Children and Adolescents With Obesity
Brief Title: Polygenic Risk Score to Predict Weight Loss Intervention in Children With Obesity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 111078-F
Record Dates: First submitted 2022-07-11; First posted 2022-07-20 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Obesity; Children
Keywords: whole exome sequencing; polygenic risk score; weight loss
MeSH Terms: conditions — Obesity; Genetic Risk Score; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — serum, WBC DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children with obesity are prone to suffering from metabolic diseases, which undoubtedly increases the burden of public health. Since obesity is a multiple gene disease, a comprehensive approach using polygenic risk scores (PRS), rather than individual genetic variant, may be a more appropriate method. The aim of the study was to establish a polygenic risk score model to assess differences to assess differences in weight loss treatment outcomes.

DETAILED DESCRIPTION:
The investigators hypothesize that obesity gene variants can predict the efficacy of weight loss intervention in obese children. The aim of the study was to establish a polygenic risk score model to assess differences to assess differences in weight loss treatment outcomes. The investigators will also analyze whether these gene variants have an effect on obesity comorbidities (hypertension, hyperlipidemia, non-alcoholic fatty liver disease, type 2 diabetes, obstructive sleep apnea, polycystic ovary syndrome, etc.). For participants with non-simple obesity, the investigators will collect their complete family history, and perform whole exome sequencing to identify possible rare disease-causing genes.

The experimental design is as follows:

Obese children and adolescent subjects will undergo a 6-month weight loss intervention program and be followed for 12-18 months. The investigators will analyze obesity and fatty liver-related genes in these adolescents using next-generation gene sequencing and/or gene chips, perform polygenic risk score analysis, and use an additive model to total the number of variant loci weighted by effect size. Whole exome gene sequencing refers to the human DNA map (hg19), and Sanger sequencing will be used to confirm the correctness of the variant site.

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years old
* Obesity definition: BMI > 95% according to the age- and gender-specific standard by National Health Institute in Taiwan
* Willing to give written informed consent

Exclusion Criteria:

* Alcohol consumption
* Major systemic diseases, including cardiopulmonary disease, renal failure, cancer, and major psychotic disorder

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Obese children and adolescents
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
weight loss | 6 month
  changes of weight and/or BMI z score
obesity severity | 1 month
  BMI z score/BMI percentile
fatty liver | 1 month
  quantification by liver ultrasound/Fibroscan

SECONDARY OUTCOMES:
hyperlipidemia | 1 month
  including triglyceride, HDL cholesterol, total cholesterol
hypertension | 1 month
  systolic and diastolic blood pressure
fasting glucose | 1 month
  hyperglycemia
HbA1c | 1 month
  hyperglycemia
2 hours glucose tolerance test | 1 month
  hyperglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Cheng Lin,, M.D., Ph.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cali AM, Caprio S. Obesity in children and adolescents. J Clin Endocrinol Metab. 2008 Nov;93(11 Suppl 1):S31-6. doi: 10.1210/jc.2008-1363. PMID 18987268
- [Background] El-Sayed Moustafa JS, Froguel P. From obesity genetics to the future of personalized obesity therapy. Nat Rev Endocrinol. 2013 Jul;9(7):402-13. doi: 10.1038/nrendo.2013.57. Epub 2013 Mar 26. PMID 23529041
- [Background] Bradfield JP, Taal HR, Timpson NJ, Scherag A, Lecoeur C, Warrington NM, Hypponen E, Holst C, Valcarcel B, Thiering E, Salem RM, Schumacher FR, Cousminer DL, Sleiman PM, Zhao J, Berkowitz RI, Vimaleswaran KS, Jarick I, Pennell CE, Evans DM, St Pourcain B, Berry DJ, Mook-Kanamori DO, Hofman A, Rivadeneira F, Uitterlinden AG, van Duijn CM, van der Valk RJ, de Jongste JC, Postma DS, Boomsma DI, Gauderman WJ, Hassanein MT, Lindgren CM, Magi R, Boreham CA, Neville CE, Moreno LA, Elliott P, Pouta A, Hartikainen AL, Li M, Raitakari O, Lehtimaki T, Eriksson JG, Palotie A, Dallongeville J, Das S, Deloukas P, McMahon G, Ring SM, Kemp JP, Buxton JL, Blakemore AI, Bustamante M, Guxens M, Hirschhorn JN, Gillman MW, Kreiner-Moller E, Bisgaard H, Gilliland FD, Heinrich J, Wheeler E, Barroso I, O'Rahilly S, Meirhaeghe A, Sorensen TI, Power C, Palmer LJ, Hinney A, Widen E, Farooqi IS, McCarthy MI, Froguel P, Meyre D, Hebebrand J, Jarvelin MR, Jaddoe VW, Smith GD, Hakonarson H, Grant SF; Early Growth Genetics Consortium. A genome-wide association meta-analysis identifies new childhood obesity loci. Nat Genet. 2012 May;44(5):526-31. doi: 10.1038/ng.2247. PMID 22484627
- [Background] Gurdasani D, Barroso I, Zeggini E, Sandhu MS. Genomics of disease risk in globally diverse populations. Nat Rev Genet. 2019 Sep;20(9):520-535. doi: 10.1038/s41576-019-0144-0. Epub 2019 Jun 24. PMID 31235872
- [Background] Holzapfel C, Sag S, Graf-Schindler J, Fischer M, Drabsch T, Illig T, Grallert H, Stecher L, Strack C, Caterson ID, Jebb SA, Hauner H, Baessler A. Association between Single Nucleotide Polymorphisms and Weight Reduction in Behavioural Interventions-A Pooled Analysis. Nutrients. 2021 Mar 2;13(3):819. doi: 10.3390/nu13030819. PMID 33801339
- [Background] Heitkamp M, Siegrist M, Molnos S, Brandmaier S, Wahl S, Langhof H, Grallert H, Halle M. Obesity Genes and Weight Loss During Lifestyle Intervention in Children With Obesity. JAMA Pediatr. 2021 Jan 1;175(1):e205142. doi: 10.1001/jamapediatrics.2020.5142. Epub 2021 Jan 4. PMID 33315090
- [Background] Herrera BM, Lindgren CM. The genetics of obesity. Curr Diab Rep. 2010 Dec;10(6):498-505. doi: 10.1007/s11892-010-0153-z. PMID 20931363
- [Background] Walley AJ, Asher JE, Froguel P. The genetic contribution to non-syndromic human obesity. Nat Rev Genet. 2009 Jul;10(7):431-42. doi: 10.1038/nrg2594. PMID 19506576
- [Background] Wand H, Lambert SA, Tamburro C, Iacocca MA, O'Sullivan JW, Sillari C, Kullo IJ, Rowley R, Dron JS, Brockman D, Venner E, McCarthy MI, Antoniou AC, Easton DF, Hegele RA, Khera AV, Chatterjee N, Kooperberg C, Edwards K, Vlessis K, Kinnear K, Danesh JN, Parkinson H, Ramos EM, Roberts MC, Ormond KE, Khoury MJ, Janssens ACJW, Goddard KAB, Kraft P, MacArthur JAL, Inouye M, Wojcik GL. Improving reporting standards for polygenic scores in risk prediction studies. Nature. 2021 Mar;591(7849):211-219. doi: 10.1038/s41586-021-03243-6. Epub 2021 Mar 10. PMID 33692554
- [Background] Eddowes PJ, Sasso M, Allison M, Tsochatzis E, Anstee QM, Sheridan D, Guha IN, Cobbold JF, Deeks JJ, Paradis V, Bedossa P, Newsome PN. Accuracy of FibroScan Controlled Attenuation Parameter and Liver Stiffness Measurement in Assessing Steatosis and Fibrosis in Patients With Nonalcoholic Fatty Liver Disease. Gastroenterology. 2019 May;156(6):1717-1730. doi: 10.1053/j.gastro.2019.01.042. Epub 2019 Jan 25. PMID 30689971
- [Background] Khera AV, Chaffin M, Wade KH, Zahid S, Brancale J, Xia R, Distefano M, Senol-Cosar O, Haas ME, Bick A, Aragam KG, Lander ES, Smith GD, Mason-Suares H, Fornage M, Lebo M, Timpson NJ, Kaplan LM, Kathiresan S. Polygenic Prediction of Weight and Obesity Trajectories from Birth to Adulthood. Cell. 2019 Apr 18;177(3):587-596.e9. doi: 10.1016/j.cell.2019.03.028. PMID 31002795
- [Background] Ford AL, Hunt LP, Cooper A, Shield JP. What reduction in BMI SDS is required in obese adolescents to improve body composition and cardiometabolic health? Arch Dis Child. 2010 Apr;95(4):256-61. doi: 10.1136/adc.2009.165340. Epub 2009 Dec 4. PMID 19966092
- [Background] Sun C, Kovacs P, Guiu-Jurado E. Genetics of Obesity in East Asians. Front Genet. 2020 Oct 20;11:575049. doi: 10.3389/fgene.2020.575049. eCollection 2020. PMID 33193685
- See also: From obesity genetics to the future of personalized obesity therapy — https://doi.org/10.1038/nrendo.2013.57
- See also: A genome-wide association meta-analysis identifies new childhood obesity loci — https://doi.org/10.1038/ng.2247
- See also: Genomics of disease risk in globally diverse populations — https://doi.org/10.1038/s41576-019-0144-0
- See also: The genetics of obesity — https://doi.org/10.1007/s11892-010-0153-z
- See also: The genetic contribution to non-syndromic human obesity — https://doi.org/10.1038/nrg2594
- See also: Improving reporting standards for polygenic scores in risk prediction studies — https://doi.org/10.1038/s41586-021-03243-6
- See also: Accuracy of FibroScan Controlled Attenuation Parameter and Liver Stiffness Measurement in Assessing Steatosis and Fibrosis in Patients With Nonalcoholic Fatty Liver Disease. Gastroenterology — https://doi.org/10.1053/j.gastro.2019.01.042
- See also: Polygenic Prediction of Weight and Obesity Trajectories from Birth to Adulthood — https://doi.org/10.1016/j.cell.2019.03.028
- See also: What reduction in BMI SDS is required in obese adolescents to improve body composition and cardiometabolic health? — https://doi.org/10.1136/adc.2009.165340
- See also: Genetics of Obesity in East Asians — https://doi.org/10.3389/fgene.2020.575049